CLINICAL TRIAL: NCT05107869
Title: Effect of Plasma Ceramides on Peripheral Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Julie K. Freed, Associate Professor, Director of Clinical Research, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 00041566
Record Dates: First submitted 2021-10-04; First posted 2021-11-04 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Vascular Disease; Lipid Disorder; Endothelial Dysfunction
Keywords: Ceramide; Endothelium
MeSH Terms: conditions — Peripheral Vascular Diseases; Lipid Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medium Chain Fatty Acid High Fat Meal (Active Comparator): This arm will assess the effect of increased plasma ceramide on peripheral microvascular function after consuming a medium chain fatty acid high fat meal.
  Interventions: Other: High Saturated Fat
- Long Chain Fatty Acid High Fat Meal (Experimental): This arm will assess the effect of increased plasma ceramide on peripheral microvascular function after consuming a long chain fatty acid high fat meal.
  Interventions: Other: High Saturated Fat

INTERVENTIONS:
Other: High Saturated Fat — High saturated fat meal

SUMMARY:
The goal of this clinical trial is to determine the effect of elevated plasma ceramides on peripheral vascular function. Subjects will consume a high fat meal consisting of long chain fatty acids (to increase plasma ceramides) or medium chain fatty acids (control). Subjects' vascular function will be assessed with laser Doppler flowmetry to measure their artery function and with the CytoCam device to assess their peripheral microvascular endothelial function.

DETAILED DESCRIPTION:
Purpose: The overarching goal of this project is to correlate the effects of plasma ceramide with human in vivo vascular function.

Formulation of Research Questions: Following decades of decline in mortality, death due to heart disease is increasing, and remains the #1 cause of death in the United States. Although acute ischemic events are typically due to obstructive plaque within the coronary conduit arteries, strong evidence suggests that dysfunction within the coronary microvasculature is a more powerful predictor of major adverse cardiac events (MACE) than severity of atherosclerosis1. The coronary microvasculature likely also contributes to other forms of cardiovascular disease including heart failure with preserved ejection fraction (HFpEF)2. While assessment of the coronary microvasculature is highly invasive and expensive, interrogation of the peripheral microvasculature offers a more feasible approach. Recent studies have concluded that peripheral microvascular dysfunction mirrors the functional status of the coronary microvasculature3. Further, impaired peripheral microvascular function is associated with increased risk of MACE in patients with stable coronary artery disease (CAD), suggesting that the microvasculature plays a critical role in the pathogenesis of heart disease4.

Elevated plasma ceramides are also associated with risk of MACE in otherwise healthy individuals5 as well as in heart failure both with and without reduced ejection fraction (HFrEF and HFpEF, respectively)6. Recently it was shown that ceramide levels are increased in patients with early CAD that also exhibit impaired coronary microvascular endothelial dysfunction7. Using an in vitro model, the investigators have previously shown that exposure to exogenous ceramide causes microvascular endothelial dysfunction in arterioles from healthy individuals8. However the effect of ceramide on human in vivo peripheral microvascular function represents a critical knowledge gap that needs to be addressed. Increased plasma ceramide may evoke peripheral in vivo microvascular dysfunction that mirrors that of the coronary microvasculature thus providing a less invasive means to assess future cardiovascular risk.

Hypothesis: Following a single high-fat meal, increases in plasma ceramides will correlate with a reduction in peripheral large and small vascular function in the intact human adult.

At Adult TRU:

1. Patient arrives at the Adult Translational Unit (ATRU) and checks in with the nurse at the front desk.
2. TRU nurse informs study team that the subject has arrived.
3. Dr. Freed or study team member consents the subject.
4. Once the subject completes the consent form, the nurse brings them to the patient room.

   1. If the subject is female, they are required to take a pregnancy test.
   2. The nurse completes the pregnancy test and gives the results to the study team member.
   3. The nurse takes baseline vital signs (height, weight, blood pressure, heart rate).
5. Baseline testing begins: (time 0)

   1. Baseline blood draw (10mL) to measure plasma ceramide levels.
   2. Baseline flow-mediated dilation (FMD) and reactive hyperemia measurements
   3. Baseline cytocam assessment
6. High-fat meal: Subjects will be given one high-fat meal by the ATRU dietitian to be ingested within 20 minutes.
7. 2-hour timepoint testing: (time 2)

   1. Blood draw (10mL) at 2hrs post initiation of high-fat meal to measure ceramide levels
   2. FMD and reactive hyperemia measurements
8. 4-hour timepoint testing: (time 4)

   1. Blood draw (10mL) at 4hrs post initiation of high-fat meal to measure ceramide levels
   2. FMD and reactive hyperemia measurements
   3. 4-hour cytocam assessment
9. After the study is completed, the patient remains in the exam room for 30 min under nurse observation

   1. During this time, vital signs are assessed by the nurse
   2. The patient may order food off the Froedtert menu

Flow-Mediated Dilation/Reactive Hyperemia Protocol Flow mediated dilation (FMD) and blood flow velocity will be assessed using a portable ultrasound machine with a 13 mHz probe. All images will be continuously captured onto using the Vascular Imager (Medical Imaging, Iowa City, IA) software. Artery diameter will automatically be measured using the boarder sensing function in the Brachial Analyzer (Medical Imaging) software.

After the subjects have rested in the supine position for 15 minutes their arm will be abducted ~80° with the pneumatic cuff placed on their forearm. Baseline brachial artery diameter and blood flow velocity through the artery will be measured 3 cm proximal to the antecubital fossa. The ultrasound probe will be positioned at 90° to the vessel to visualize anterior and posterior lumen-intimal interfaces. After baseline images have been captured, the pneumatic cuff will be inflated to 225 mmHg for 5 minutes to occlude blood flow to the lower leg or forearm. Immediately after cuff release, the increased blood flow velocity due to the reactive hyperemia response will be measured. To assess vasodilation, images will be captured at a rate of 10 images/second for 3 minutes after cuff release.

Cytocam Assessment for Microvascular Function Approximately 10 images will be taken to establish a baseline. The study team will administer 1% acetylcholine (via Q-tip, liquid dropper or gauze) under the tongue for 1 minute. The CytoCam is reinserted to take approximately 10 more images. The patient will be allowed 30 minutes to rest while the nurse retakes vital signs. After 30 minutes, a new set of approximately 10 baseline images are taken. The study team will administer a nitroglycerin tablet (0.3mg) under the tongue. Once the tablet dissolves the CytoCam will be reinserted to image the vessels (approximately 10 images) after 2-3 minutes following tablet administration.

ELIGIBILITY:
Inclusion Criteria:

1. Health adults aged 18-40 years
2. English-speaking only
3. Not pregnant

Exclusion Criteria:

1. Healthy individuals under 18 years or over 40 years of age
2. Non-English speaking
3. Pregnant individuals
4. Heart rate <60 or >100
5. Systolic blood pressure <100 or >160
6. Subjects with visible open sores or wounds in mouth
7. Lactose intolerant or allergy to dairy products
8. Diabetes Mellitus
9. Coronary Artery Disease
10. High blood pressure
11. High cholesterol
12. Heart failure
13. Current tobacco use
14. Chemotherapy within the last 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Cardiovascular Conductance | 6 hours
  Use laser Doppler flowmetry to measure blood flow
Endothelial-Dependent Total Vessel Density | 6 hours
  Use a microscope (CytoCam) to look at blood vessels

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Freed JK, Beyer AM, LoGiudice JA, Hockenberry JC, Gutterman DD. Ceramide changes the mediator of flow-induced vasodilation from nitric oxide to hydrogen peroxide in the human microcirculation. Circ Res. 2014 Aug 15;115(5):525-32. doi: 10.1161/CIRCRESAHA.115.303881. Epub 2014 Jun 11. PMID 24920698
- [Background] Akhiyat N, Vasile V, Ahmad A, Sara JD, Nardi V, Lerman LO, Jaffe A, Lerman A. Plasma Ceramide Levels Are Elevated in Patients With Early Coronary Atherosclerosis and Endothelial Dysfunction. J Am Heart Assoc. 2022 Apr 5;11(7):e022852. doi: 10.1161/JAHA.121.022852. Epub 2022 Mar 18. PMID 35301857
- [Background] Lemaitre RN, Jensen PN, Hoofnagle A, McKnight B, Fretts AM, King IB, Siscovick DS, Psaty BM, Heckbert SR, Mozaffarian D, Sotoodehnia N. Plasma Ceramides and Sphingomyelins in Relation to Heart Failure Risk. Circ Heart Fail. 2019 Jul;12(7):e005708. doi: 10.1161/CIRCHEARTFAILURE.118.005708. Epub 2019 Jul 12. PMID 31296099
- [Background] Havulinna AS, Sysi-Aho M, Hilvo M, Kauhanen D, Hurme R, Ekroos K, Salomaa V, Laaksonen R. Circulating Ceramides Predict Cardiovascular Outcomes in the Population-Based FINRISK 2002 Cohort. Arterioscler Thromb Vasc Biol. 2016 Dec;36(12):2424-2430. doi: 10.1161/ATVBAHA.116.307497. Epub 2016 Oct 20. PMID 27765765
- [Background] Al-Badri A, Kim JH, Liu C, Mehta PK, Quyyumi AA. Peripheral Microvascular Function Reflects Coronary Vascular Function. Arterioscler Thromb Vasc Biol. 2019 Jul;39(7):1492-1500. doi: 10.1161/ATVBAHA.119.312378. Epub 2019 Apr 25. PMID 31018659
- [Background] Paulus WJ, Tschope C. A novel paradigm for heart failure with preserved ejection fraction: comorbidities drive myocardial dysfunction and remodeling through coronary microvascular endothelial inflammation. J Am Coll Cardiol. 2013 Jul 23;62(4):263-71. doi: 10.1016/j.jacc.2013.02.092. Epub 2013 May 15. PMID 23684677
- [Background] van de Hoef TP, van Lavieren MA, Damman P, Delewi R, Piek MA, Chamuleau SA, Voskuil M, Henriques JP, Koch KT, de Winter RJ, Spaan JA, Siebes M, Tijssen JG, Meuwissen M, Piek JJ. Physiological basis and long-term clinical outcome of discordance between fractional flow reserve and coronary flow velocity reserve in coronary stenoses of intermediate severity. Circ Cardiovasc Interv. 2014 Jun;7(3):301-11. doi: 10.1161/CIRCINTERVENTIONS.113.001049. Epub 2014 Apr 29. PMID 24782198